CLINICAL TRIAL: NCT04290416
Title: Human Single Neuron Recordings in Epilepsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Birmingham (Other)
Collaborators: European Commission (Other); Queen Elizabeth Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG_15-074
Record Dates: First submitted 2019-12-18; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy; Memory
MeSH Terms: conditions — Epilepsy

ARMS (1):
- Microwire electrodes (Experimental): Activity of individual neurons will be recorded via microwire contacts. These microwire electrodes do not interfere with the macrowire clinical recordings.
  Interventions: Diagnostic Test: Microwire electrodes

INTERVENTIONS:
Diagnostic Test: Microwire electrodes

SUMMARY:
This study uses single neuron recordings in pre-surgical epilepsy patients to uncover the neural mechanisms underlying memory formation and retrieval. A secondary aim is to improve diagnostic tools to identify epileptogenic tissue.

ELIGIBILITY:
Inclusion Criteria:

* Interest in participation.
* Temporal lobe epilepsy that is clinically being investigated with implantations of depth electrodes as part of the pre-surgical epilepsy monitoring.
* Cognitive/language skills sufficient to follow experimental instruction and maintain focus on the experiment.

Exclusion Criteria:

* Patient does not want to participate.
* Extra-temporal epilepsy, or electrode implantation strategy that does not allow the use of micro-macrowire electrodes.
* Cognitive/language skills insufficient to follow experimental instruction and maintain focus on the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-02-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Single unit recordings | 14 days (patient in hospital for this length of time)
  Activity of individual neurons will be recorded via micro wire electrodes

SECONDARY OUTCOMES:
Intracranial electroencephalogram (iEEG) | 14 days (patient in hospital for this length of time)
  Secondary outcome measures will be iEEG signals recorded with the macro electrodes, such as:
  * Event-related potentials
  * EEG power and phase of Theta oscillations
  * EEG power and phase of Alpha/Beta oscillations
  * EEG power and phase of Gamma oscillations
  * EEG power of High Frequency Oscillations (>80 Hz)
Behavioural response data | 14 days (patient in hospital for this length of time)
  Laptop button presses and corresponding response times will be recorded in MATLAB and presentation file formats. This is acquired at patient's bedside during hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hanslmayr, PhD, Principal Investigator — University of Birmingham
Locations (1):
- Queen Elizabeth UHB Hospital, Birmingham, West Midlands, United Kingdom